CLINICAL TRIAL: NCT07181538
Title: Phase 1 Study to Evaluate the Pharmacokinetics and the Safety After Administration of "JLP-2302" and "JP-1366" in Healthy Volunteers
Brief Title: Phase 1 Study of JLP-2302 and JP-1366: PK and Safety in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JP-1366-110
Record Dates: First submitted 2025-08-29; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: pharmacokinetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JLP-2302 and JP-1366 crossover (Experimental)
  Interventions: Drug: JLP-2302; Drug: JP-1366
- JP-1366 and JLP-2302 crossover (Active Comparator)
  Interventions: Drug: JLP-2302; Drug: JP-1366

INTERVENTIONS:
Drug: JLP-2302 — taking JLP-2302
Drug: JP-1366 — taking JP-1366

SUMMARY:
This study aims to evaluate the pharmacokinetics and the safety after administration of "JLP-2302" and "JP-1366" in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a body mass index (BMI) between 18.0 and 30.0 kg/m²
* Subjects without any clinically significant congenital or chronic disease, and with no pathological findings based on medical examination
* Subjects who agree to use a medically acceptable method of contraception*

Exclusion Criteria:

* Subjects who have taken enzyme-inducing or -inhibiting drugs
* Subjects who have participated in a bioequivalence or other clinical trial and received an investigational product within 6 months prior to the first dose
* Subjects with a history of gastrointestinal surgery that may affect drug absorption
* Subjects with a clinically significant history of psychiatric illness
* Female subjects who are pregnant, suspected of being pregnant, or currently breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve(AUCt) | Pre-dose on Day 1 and on Days 2 post-dose
Peak Plasma Concentration (Cmax) | Pre-dose on Day 1 and on Days 2 post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No